CLINICAL TRIAL: NCT05358496
Title: Study of Neutrophils and Circulating Platelets in Correlation With the Activity of T Lymphocytes in Patients With NAFLD (Nonalcoholic Fatty Liver Disease)
Acronym: NAFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Clara Balsano, Full Professor, University of L'Aquila
Other Study IDs: 31869
Record Dates: First submitted 2021-09-29; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: NAFLD- Non Alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD cohort
  Interventions: Diagnostic Test: Data collection
- Validation cohort
  Interventions: Diagnostic Test: Data collection

INTERVENTIONS:
Diagnostic Test: Data collection — Clinical data collection

SUMMARY:
The aim of the study is to define the relationship between neutrophils, platelets and the activity of T lymphocytes in patients with NAFLD (nonalcoholic fatty liver disease).

This study may predict, in the course of hepatic steatosis, specific phenotypic patterns expressed by PMNs and circulating platelets to evaluate their role in disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* No alcoholic abuse
* Hepatic steatosis diagnosticated by abdominal ultrasound
* Negative hepatitis B and C tests
* No history of hepatic cirrhosis

Exclusion Criteria:

* Under 18
* History of alcoholic abuse
* Positive serology for hepatitis B or C
* History of hepatic cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Italian caucasian patients over 18 years old with NAFLD diagnosis
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
IL-8(interleukin 8) | 12 months
Morphology of Circulating Platelets in healthy donors, NAFL, and NASH patients wondering how they may drive and modulate the activity of T cells in this disease | 12 months
Platelets count in healthy donors, NAFL, and NASH patients | 12 months
number of Neutrophilis | 12 months
Morphology of Neutrophilis | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clara Balsano, L’Aquila, Italy/L'Aquila, Italy